CLINICAL TRIAL: NCT01510899
Title: A Multiple Center, Open-label, Single Dose, Parallel-group Study to Investigate the Effect of Renal Impairment on the Pharmacokinetics of RO4917838
Brief Title: A Study on the Effect of Renal Impairment on the Pharmacokinetics of RO4917838
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: BP25261
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

ARMS (2):
- Healthy Subjects Arm (Experimental)
  Interventions: Drug: RO4917838
- Renal Impaired Subjects Arm (Experimental)
  Interventions: Drug: RO4917838

INTERVENTIONS:
Drug: RO4917838 — Single dose of RO4917838
  Arms: Renal Impaired Subjects Arm
Drug: RO4917838 — Single dose of RO4917838
  Arms: Healthy Subjects Arm

SUMMARY:
This open-label, single-dose, parallel-group study will investigate the pharmacokinetics and safety of RO4917838 in healthy and renal impaired subjects. Subjects will receive a single dose of RO4917838.

ELIGIBILITY:
Inclusion Criteria:

General criteria

* Body mass index (BMI) between 18 and 32 kg/m2

Criteria applying to renal impaired subjects

* Adult subjects, 18-65 years of age
* Part 1: Subjects with end stage renal disease (ESRD), not on dialysis
* Part 2: Subjects with severe, moderate or mild renal impairment
* Stable renal function

Criteria applying to healthy subjects

* Adult subjects, 18-70 years of age

Exclusion Criteria:

General criteria

* Any condition or disease (other than renal impairment for the renal impaired subjects only) that would render the subject unsuitable for the study, or would place the subject at undue risk
* Any condition which could relapse during or immediately after the study
* History of alcohol or drug abuse

Criteria applying to renal impaired subjects

* Evidence of unstable clinically significant disease other than renal impairment
* Clinically significant liver disease
* Any other major illness (with the exception of renal impairment) within 4 weeks prior to study start

Criteria applying to healthy subjects

* History of any clinically significant disease (e.g., cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic disease)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under concentration time curve of RO4917838 | Days 1-16

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Rennes, France
- Moscow, Russia